CLINICAL TRIAL: NCT05296239
Title: Social Assistive Robot Interface for People With Alzheimers and Other Dementias to Aid in Care Management
Brief Title: SimpleC Wellness Platform With Social Robot Interaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SimpleC, LLC (Industry)
Collaborators: University of Georgia (Other); Advanced Medical Electronics (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 7645C
Record Dates: First submitted 2022-02-23; First posted 2022-03-25 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Engagement, Patient; Mood; Quality of Life; Aging; Mild Cognitive Impairment; Cognitive Impairment; Dementia
Keywords: At risk; Diagnosis
MeSH Terms: conditions — Patient Participation; Cognitive Dysfunction; Dementia; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SimpleC Wellness Platform with Social Robot Interaction (Experimental)
  Interventions: Other: SimpleC Wellness Platform with Social Robot Interaction

INTERVENTIONS:
Other: SimpleC Wellness Platform with Social Robot Interaction — Once respondents enroll, they will receive the SimpleC Wellness Platform, including introduction training on the SAR system. During the study period, participants and others will receive instructions for the SAR system and use it as part of scheduled interactions, which includes interactions as part of the general schedule. In the third week, the social robot will be installed, and staff trained in group sessions as available. Participants may use the full SAR system as they are willing.
  Interactions specific to the virtual and physical robot include notifications to join activities as per community schedule as well as trivia.

SUMMARY:
This implementation study will be conducted to test a Socially-Assistive Robot (SAR) system for residents in an Assisted Living environment. The goal of the SAR system is to enhance social engagement and connectedness. The system engages residents via robot-facilitated activities such as trivia and reminder and is integrated with the SimpleC Wellness Platform.

DETAILED DESCRIPTION:
This is a 3-week mixed-method study to assess the installation procedure, assess user first impressions, develop training, assess user materials, and identify any barriers and concerns during implementation. New features and design will be validated.

Research questions include:

* How should the SAR system be introduced to the users and their environment?
* What are facilitators and barriers to implementation?
* Will users accept the SAR system in their environment?
* What are facilitators and barriers to SAR system acceptance?
* What are the desired parameters that the SAR system should have?

  * What social behaviors do users expect?
  * What tasks would be acceptable that the SAR system tablet do?
  * How should the SAR system's perception, competence, and awareness be presented to users?
  * What is most valuable to users and why?
* If the answer depends, then what does it depend on (user, task, environment)?

Sample: Thirty individuals will participate: 10 residents, 10 family, and 10 staff. Enrollment will stop when reaching saturation.

Procedure: The research will follow established procedures for recruitment, screening, and assessment. Participants will provide informed consent, which will be followed by a baseline assessment. Participants will be screened to ascertain inclusion and exclusion criteria. Residents and Senior Housing Community will receive the new SAR system, which includes a virtual robot and physical social robot. At the beginning of the study, enrolled residents will receive a tablet with a personalized profile, wellness programs, and virtual robot using the standard SimpleC enrollment process. Installation will be followed by training. Residents and family will be invited to personalize residents' profile and programming. One social robot will be implement for the whole community. Participants will engage with the SAR system as they are willing. All staff, residents, and family will be invited to use the SAR system, independent of study participation status. At the end of the study, assessments will be administered, which is followed by a brief interview.

ELIGIBILITY:
Inclusion Criteria:

* All: Fluent in English
* Resident: 50 years and older
* Resident: lives in Assisted Living Community
* Resident: MMSE score of 13 or higher
* Family member: 18 years and older
* Family member: family or friend of resident
* Family member: no diagnosis of dementia or related disorder
* Staff: 18 years and older
* Staff: works for the Senior Housing Community

Exclusion Criteria:

* All: pregnant
* Resident: Expecting to move during the study
* Resident: Both legally deaf and blind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Facilitators to successful implementation | 3 weeks
  Identified factors that facilitate successful implementation (e.g., WiFi, environmental set up, user perceptions) as derived from analysis of: [interview, observational notes, usage data]
Barriers to successful implementation | 3 weeks
  Identified factors that are barriers to implementation (e.g., WiFi, environmental set up, user perceptions) as derived from: [interview, observational notes, usage data]

SECONDARY OUTCOMES:
Technology Acceptance Model Questionnaire. A 12-item scale with high scores indicating higher acceptance. | 3 weeks
  [Questionnaires] Assessment of users' perceived ease of use, usefulness, and satisfaction of using the technology.
Technology acceptance and adoption | 3 weeks
  [Interview] Assessment of users acceptance and adoption ease of use, usefulness, and satisfaction of using the technology.
Robotic Social Attributes Scale (RoSAS). An 18-item scale with high scores indicating positive attitudes for dimensions of warmth and competency and a negative attitude for dimension of discomfort. | 3 weeks
  [Questionnaire] Perception and judgment of Social Assistive Robot social attributes on 3 dimensions: Warmth, competency, and discomfort
Robot Social Attributes | 3 weeks
  [Interview] Social Assistive Robot social attributes are identified (e.g., friendliness, competency, etc)
Usability and usefulness | 3 weeks
  Identified factors that indicate the ease of use and usefulness for different tasks as derived from analysis of: [Interview, usage data]
Conversation quality | 3 weeks
  [Interview] User perceptions on the usefulness and ease of use in conversing with the technology.
Value proposition/Economic Impact | 3 weeks
  [Interview] Discussions with facility staff and key decision makers to understand the value of the technology in providing social interaction and reminders to their residents.
Requirements | 3 weeks
  Identified requirements for design, training, and communication as derived from analysis of: [Interview, observations]
Affect | 3 weeks
  [Interview] Feelings of enjoyment, satisfaction, when using the technology
Guilt Scale. A 4-point scale with higher score indicating higher guilt. | 3 weeks
  [Questionnaire] Family caregiver feelings of guilt.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Adams, PhD, Principal Investigator — SimpleC, LLC; Jenay Beer, PhD, Principal Investigator — jenay.beer@uga.edu
Locations (2):
- United States (2):
  - University of Georgia, Athens, Georgia
  - SimpleC, LLC, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No